CLINICAL TRIAL: NCT06577467
Title: Cross-Sectional Evaluation of Persistence of SARS-CoV-2 Remnants After Recovery From Acute Infection
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002067; 002067-N
Record Dates: First submitted 2024-08-28; First posted 2024-08-29 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11-25

CONDITIONS: PASC Post Acute Sequelae of COVID-19
Keywords: PASC; COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuro-PASC: 1.<TAB>Neurologic and neuropsychiatric complaint is the primary clinical issue. 2.<TAB>Neuro-PASC clinical symptom burden is moderate or greater.3.<TAB>Other PASC complications, such as pulmonary, cardiovascular, or gastrointestinal symptoms, are not prominent case features.
- Recovered volunteers: 1.<TAB>Reports no ongoing or new health issues attributable to a SARS-CoV-2 infection2.<TAB>Overall clinical symptoms burden is no greater than mild3.<TAB>No clinically substantial comorbid medical or psychiatric conditions

SUMMARY:
Background:

SARS-CoV-2 is the virus that causes COVID-19. Some people who recover from COVID-19 have symptoms that last long after the active infection ends. This is called long COVID. Sometimes, long COVID can affect the nerves and cause problems with sleep, thinking, the senses, and movement. Researchers want to find out whether people with long COVID have retained inactive remnants of SARS-CoV-2 in their bodies.

Objective:

To collect tissue samples to see if people with long COVID have remnants of SARS-CoV-2 in their bodies.

Eligibility:

People 18 years or older who have recovered from COVID-19, both with and without neurologic symptoms.

Design:

Participants will have 2 to 4 inpatient or outpatient visits over 4 months. Each visit will last 4 to 5 days.

Participants will be screened to make sure it is safe to collect tissue samples from their body. They will have a physical and dental exam. They will have imaging scans and a test of their heart function. They will complete questionnaires about their health. They will give blood, urine, saliva, and stool samples. Their sense of taste and smell will be tested.

Tissue samples will be taken from the digestive tract, lungs, colon, skin, muscle, lymph nodes, nasal passages, and mouth. Participants may be numbed or sedated for some of the procedures.

Swabs will be used to collect cells from inside the mouth and nose.

Participants will undergo lumbar puncture. A thin needle will be inserted into their lower back to draw out a sample of the fluid around their spinal cord.

Participants will have follow-up phone calls after each clinic visit.

DETAILED DESCRIPTION:
Study Description:

It has been demonstrated that remnants of the SARS-CoV-2 virus remain after the resolution of the acute infective period. It is not known if these viral remnants interact with host tissues in the development and maintenance of the Post-Acute Sequelae of COVID-19 (PASC)/Long COVID. Better understanding of how to recover and characterize SARS-CoV-2 viral remnants from humans is a valuable first step in understanding the health impact that they may have on humans. This study will focus on the recovery and characterization of SARS-CoV-2 remnants from multiple organ sites of individual volunteers with persistent neurological complications from SARS-CoV-2 (Neuro-PASC) and volunteers those who have recovered from a SARS-CoV-2 infection (RV).

Objectives:

* Primary Objective:

  --To determine where remnants of SARS-CoV-2 virus can be recovered in persons with neuro-PASC and RVs.
* Secondary Objectives:

  * To characterize the biochemical nature of SARS-CoV-2 recovered viral remnants (e.g. proteins, nucleic acids).
  * To determine if there are quantitative differences in recovered SARS-CoV-2 proteins between neuro-PASC and RV participants.
  * To determine if there are quantitative differences in recovered SARS-CoV-2 nucleic acids between neuro-PASC and RV participants.

Endpoints:

This is an exploratory cross-sectional protocol to determine whether the presence or absence of viral remnants can be detected in a range of human tissues. Hence, tissue-specific detection of viral remnants is the primary end point. Secondary endpoints will characterize and quantify the recovered remnants to allow group comparisons between neuro-PASC and RV participants.

ELIGIBILITY:
* INCLUSION CRITERIA:

Recovered Volunteers (RV): Six healthy persons who have recovered from an acute SARS-CoV-2 infection.

Inclusion criteria:

* Participants 18 and older
* Ability to provide informed consent
* Completed participation in Phase B of Protocol 000089
* Met 000089 Inclusion criteria for Mild to Moderate COVID-19 without PASC symptoms:

  * Licensed Independent Practitioner documentation of a stable state of general well health and physical function prior to contracting SARS-CoV-2. This may include medical records, correspondence letters, or information gathered from telephone calls with study personnel.
  * A self-reported illness narrative of recovery to prior health after a SARS/CoV2 infection.
  * Laboratory documentation of a positive COVID-19 PCR, NAA, or other EUA approved test to confirm active COVID infection at the time of the SARS-CoV-2 infection. Participants with positive home tests during Phase A will be required to have a positive anti-SARS nucleocapsid antibody test.
  * Meets WHO Clinical Progression Scale of 2 - 6:

    2: Ambulatory; symptomatic, independent

    3: Ambulatory; symptomatic, assistance needed

    4: Hospitalized; no oxygen therapy

    5: Hospitalized; oxygen by mask or nasal prongs

    6: Hospitalized; oxygen by non-invasive ventilation or high flow oxygen
  * Functional Criteria: No substantial symptom severity as determined using SF-36v2: score of >=85 physical function subscale, and >=85 on role physical subscale, and >=85 on social function subscale.
* Determined to be a Healthy Comparator by the 000089 Case Adjudication Committee
* Does not have an active SARS-CoV-2 infection. The protocol will conform with NIH CC standards for documenting a participant does not have active SARS-CoV-2 infection. This may include screening interviews and/or testing. Testing may be repeated with each admission. Participants may be rescreened 6 weeks after acute infection has resolved.

Neurologic Post-Acute Sequelae of COVID-19 Participants (Neuro-PASC):

Six persons with ongoing neurological complaints following an acute SARS-CoV-2 infection.

Inclusion criteria:

* Participants 18 and older
* Ability to provide informed consent
* Completed participation in Phase B of Protocol 000089
* Met 000089 Inclusion criteria for Mild to Moderate COVID-19 with PASC symptoms:

  * Licensed Independent Practitioner documentation of a stable state of general well health and physical function prior to contracting SARS-CoV-2. This may include medical records, correspondence letters, or information gathered from telephone calls with study personnel.
  * A self-reported illness narrative of the development of persistent PASC symptoms after recovering from a SARS-CoV-2 infection. These include symptoms such as fatigue, cognitive difficulties, orthostatic intolerance, unrefreshing sleep, neuropathic pain, mood change, and post-exertional malaise.
  * Laboratory documentation of a positive COVID-19 PCR, NAA, or other EUA approved test to confirm active COVID infection at the time of the SARS-CoV-2 infection. Participants with positive home tests during Phase A will be required to have a positive anti-SARS nucleocapsid antibody test .
  * Meets WHO Clinical Progression Scale of 2 - 6:

    2: Ambulatory; symptomatic, independent

    3: Ambulatory; symptomatic, assistance needed

    4: Hospitalized; no oxygen therapy

    5: Hospitalized; oxygen by mask or nasal prongs

    6: Hospitalized; oxygen by non-invasive ventilation or high flow oxygen
  * Functional Criteria: Substantial symptom severity as determined using SF-36v2: score of <= 70 physical function subscale, or <=50 on role physical subscale, or <=75 on social function subscale.
* Determined to have Post-Acute Sequelae of COVID-19 by the 000089 Case Adjudication Committee
* Primary PASC complaint is neurologic including:

  * Neuropathic sensations
  * Cognitive complaints
  * Postural (Orthostatic) complaints
  * Motor complaints
* Does not have an active SARS-CoV-2 infection. The protocol will conform with NIH CC standards for documenting a participant does not have active SARS-CoV-2 infection. This may include screening interviews and/or testing. Testing may be repeated with each admission. Participants may be rescreened 6 weeks after acute infection has resolved.

EXCLUSION CRITERIA:

* Current suicidal ideation
* Women who are pregnant, breastfeeding, or are within one-year post-partum.
* Current or previous malignancy. A history of malignancy that has fully resolved with surgical resection only (e.g. no chemotherapy, radiation therapy, or immunotherapy) will be allowed.
* Current systemic immunologic disorders (e.g. Type 1 diabetes, rheumatoid arthritis). Local immunological disorder (e.g. atopic dermatitis, stable autoimmune thyroid disease) and allergic disorders will be allowed.
* Current or previous long-term immune suppressive therapy. Systemic steroid use, even short-term, must not have been used within the month prior to enrollment.
* Long term use of anticoagulant or antiplatelet medications.
* Active participation in a clinical protocol (e.g. anti-inflammatory drug intervention study) which includes an intervention that may affect the results of the current study.
* Not willing to allow for research data and samples to be shared broadly with other researchers.
* Employees of NIH.
* Symptom severity that makes it impossible for the volunteer to travel to NIH for an extended inpatient evaluation
* Use of medications with a high-risk for withdrawal-related complications (i.e. long-acting opiates or benzodiazepines).
* Unwillingness to co-enroll in protocol 17-I-0122: NIAID Centralized Sequencing Protocol.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 6 neuro-PASC patients with: 1. Neurologic and neuropsychiatric complaint is the primary clinical issue. 2. Neuro-PASC clinical symptom burden is moderate or greater. 3. Other PASC complications, such as pulmonary, cardiovascular, or gastrointestinal symptoms, are not prominent case features. 6 Recovered volunteers with: 1. Reports no ongoing or new health issues attributable to a SARS-CoV-2 infection 2. Overall clinical symptoms burden is no greater than mild 3. No clinically substantial comorbid medical or psychiatric conditions
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
To determine where remnants of SARS-CoV-2 virus can be recovered in persons with neuro-PASC and RVs. | Study End
  This is an exploratory study to determine where SARS-CoV-2 viral remnants can be recovered in tissues of patients with Neuro-PASC.

SECONDARY OUTCOMES:
1.To characterize the biochemical nature of SARS-CoV-2 recovered viral remnants (e.g. proteins, nucleic acids).PASC and RV participants. | Study End
  If defective or restricted viral replication is present in the tissues, one might not detect fully replicating virus or all viral components. It is not known if SARS-CoV-2 proteins or RNA preferentially resides in particular tissue types.
2.To determine if there are quantitative differences in recovered SARS-CoV-2 proteins between neuro-PASC and RV participants. | Study End
  If defective or restricted viral replication is present in the tissues, one might not detect fully replicating virus or all viral components. It is not known if SARS-CoV-2 proteins or RNA preferentially resides in particular tissue types.
3.To determine if there are quantitative differences in recovered SARS-CoV-2 nucleic acids between neuro-PASC and RV participants. | Study End
  If defective or restricted viral replication is present in the tissues, one might not detect fully replicating virus or all viral components. It is not known if SARS-CoV-2 proteins or RNA preferentially resides in particular tissue types.

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared that underlie results in a publication.
Supporting Information: Study Protocol, ICF
Time Frame: At time of publication
Access Criteria: Creative commons-BY

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002067-N.html